CLINICAL TRIAL: NCT07268131
Title: Neoadjuvant TACE Plus Iparomlimab and Tuvonralimab （QL1706）and Adjuvant QL1706 in Resectable BCLC Stage A/B Hepatocellular Carcinoma Patients Beyond Milan Criteria: the TITAN-HCC Phase II Trial
Brief Title: TITAN-HCC: Neoadjuvant and Adjuvant QL1706 With TACE in Resectable Hepatocellular Carcinoma Beyond Milan Criteria
Acronym: TITAN-HCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-875
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE+QL1706 (Experimental): TACE+QL1706 (PD-1/CTLA-4 antibody, 7.5mg/kg, ivgtt, Q3W)
  Interventions: Combination Product: TACE+QL1706

INTERVENTIONS:
Combination Product: TACE+QL1706 — TACE+QL1706(PD-1/CTLA-4 antibody, 7.5mg/kg, ivgtt, Q3W)

SUMMARY:
This is a single-arm, single-center, prospective trial designed to evaluate the efficacy and safety of transarterial chemoembolization (TACE) combined with ipalimab/tuvonralimab (QL1706) in the peri-operative setting for resectable hepatocellular carcinoma exceeding the Milan criteria, and to explore biomarkers predictive of therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female
* Patients with histologically or pathologically confirmed hepatocellular carcinoma (HCC), or Patients meeting the clinical diagnostic criteria for hepatocellular carcinoma as defined by the American Association for the Study of Liver Diseases (AASLD)
* BCLC stage A or B hepatocellular carcinoma deemed amenable to curative-intent surgery after multidisciplinary consultation, yet exceeding Milan criteria
* Eligible for the TACE procedure predefined by the study center, with no contraindications
* Child-Pugh score ≤7
* ECOG PS ≤1
* Measurable disease per RECIST 1.1 criteria
* Life expectancy >12 weeks
* Adequate organ function meeting the following laboratory values: Hematological: Absolute neutrophil count (ANC) ≥1.5×10⁹/L Platelet count (PLT) ≥75×10⁹/L Hemoglobin (HGB) ≥90 g/L Hepatic: Total bilirubin (TBIL) ≤3× upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5×ULN Serum albumin ≥28 g/L Note: Patients may be enrolled if values stabilize after standard liver support therapy for ≥1 week, as assessed by the investigator. Renal: Serum creatinine (Cr) ≤1.5×ULN or Creatinine clearance ≥50 mL/min (calculated by Cockcroft-Gault formula) Coagulation: International normalized ratio (INR) ≤2×ULN or Activated partial thromboplastin time (APTT) ≤2×ULN
* Willing and able to provide written informed consent prior to any study-related procedures

Exclusion Criteria:

* Patients with histopathologically confirmed variant hepatocellular carcinoma (HCC) subtypes, including: Fibrolamellar hepatocellular carcinoma Sarcomatoid hepatocellular carcinoma Mixed hepatocellular-cholangiocarcinoma
* Prior local therapy targeting the index lesion(s), including but not limited to: Transarterial chemoembolization (TACE) Transarterial embolization (TAE) Transarterial radioembolization (TARE) Hepatic arterial infusion chemotherapy (HAIC) Radiofrequency ablation (RFA) Cryoablation High-intensity focused ultrasound (HIFU) Radiation therapy
* Prior systemic anti-cancer therapy for hepatocellular carcinoma, including but not limited to: Molecular targeted agents (e.g., tyrosine kinase inhibitors, anti-angiogenic drugs) Conventional chemotherapy Immunotherapy: Immune checkpoint inhibitors (e.g., PD-1/PD-L1/CTLA-4 inhibitors) Immune checkpoint agonists Cellular immunotherapy (e.g., CAR-T, NK cell therapy) Biological therapy: Cancer vaccines Cytokines (e.g., interferons, interleukins) Growth factor inhibitors
* Presence of portal vein tumor thrombus, hepatic vein or inferior vena cava tumor thrombus, or distant metastasis
* History of bleeding events within 6 months prior to initial treatment, including but not limited to: Acute hemorrhage from esophageal or gastric varices caused by portal hypertension AND/OR 6. Untreated or inadequately treated
* Clinically significant cardiovascular or cerebrovascular disease, including any of the following within 3 months prior to initial treatment: Congestive heart failure (NYHA Class ≥II) Myocardial infarction Cerebrovascular accident (stroke/TIA) Unstable arrhythmia Unstable angina OR 8. History of congenital long QT syndrome OR 9. Screening ECG showing QTc interval >500 ms (calculated by Fridericia's formula)
* Active autoimmune disease requiring systemic treatment (e.g., disease-modifying agents, corticosteroids, immunosuppressants) within 2 years prior to initial treatment, with the following exceptions: Non-systemic replacement therapies (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal/pituitary insufficiency)
* Known HIV-positive status or history of active acquired immunodeficiency syndrome (AIDS)
* History of allogeneic stem cell transplantation or solid organ transplantation
* History of other active malignancies within 5 years prior to initial treatment, except for those with negligible risk of metastasis or death (e.g., 5-year overall survival rate >90%), including: Adequately treated carcinoma in situ of the cervix Non-melanoma skin cancer Localized prostate cancer (Gleason score ≤6, treated if required) Superficial bladder cancer (Ta/Tis, non-invasive)
* Women who are pregnant or breastfeeding
* Concurrent participation in another clinical trial, unless: It is a non-interventional study (e.g., observational/registry study), OR The patient is in the follow-up phase of an interventional trial, defined as: ≥4 weeks since last dose in the prior trial, OR ≥5 half-lives of the investigational drug (whichever is shorter)
* Systemic corticosteroid (>10 mg/day prednisone or equivalent) or other immunosuppressive therapy within 2 weeks prior to initial treatment, with the following exceptions: Adrenal replacement therapy (prednisone ≤10 mg/day or equivalent) Topical, ocular, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption Short-term corticosteroid prophylaxis for hypersensitivity reactions (e.g., premedication for CT scans)
* Any clinical or laboratory abnormality or compliance issue deemed by the investigator to render the patient unsuitable for enrollment in this clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response（MPR） | Periprocedural
  In the tumor bed of the surgical resection specimen, necrotic or regressive tumor tissue ≥90 %.